CLINICAL TRIAL: NCT02071173
Title: Evaluation of ACUITY™ X4 Quadripolar Coronary Venous Leads and RELIANCE™ 4-FRONT Defibrillation Leads: NAVIGATE X4
Brief Title: Evaluation of ACUITY™ X4 Quadripolar Coronary Venous Leads and RELIANCE™ 4-FRONT Defibrillation Leads
Acronym: NAVIGATE X4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1481
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Cardiac Resynchronization Therapy

STUDY DESIGN:
Intervention Model Description: Every subject had access to two study devices and were followed as a single group.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enrolled Patients (Experimental): Subjects undergo an implant procedure to receive at least one investigational lead -- ACUITY X4 left ventricular (LV) CRT lead, RELIANCE 4-FRONT right ventricular (RV) ICD lead
  Interventions: Device: ACUITY X4 quadripolar coronary venous lead and RELIANCE 4-FRONT defibrillation lead

INTERVENTIONS:
Device: ACUITY X4 quadripolar coronary venous lead and RELIANCE 4-FRONT defibrillation lead — The ACUITY X4 leads are intended for chronic left ventricular pacing and sensing. The leads have 3 tip configuration designs (straight tip, short tip spiral, and long tip spiral), which is intended to provide choices for patients with different anatomies.
  The RELIANCE 4-FRONT leads are designed for right-side heart applications within the ventricle, atrium, and superior vena cava. It is intended for permanent sensing, pacing, and defibrillation when used with a compatible implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy defibrillator (CRT-D).
  Subjects were allowed to receive both the ACUITY X4 and RELIANCE 4-FRONT lead.
  Other Names: LV Quadripolar coronary venous lead; RV defibrillation Lead

SUMMARY:
The objective of the NAVIGATE X4 Clinical Study is to gather data to establish the safety, performance and effectiveness of the ACUITY™ X4 quadripolar coronary venous leads and the RELIANCE 4-FRONT™ ventricular defibrillation leads to satisfy FDA requirements for pre-market submission. Additionally, data from this study will be used to support post-market approval requirements for the ACUITY X4 and RELIANCE 4-FRONT leads.

ELIGIBILITY:
Inclusion Criteria:

Subjects indicated for a CRT-D that fulfill one of the following 5 criteria[1]:

1. Subject with left ventricular ejection fraction (LVEF) less than or equal to 35%, sinus rhythm, left bundle branch block (LBBB) with a QRS duration greater than or equal to 150 ms, and a NYHA class II, III or ambulatory IV symptoms on Guideline-Directed Medical Therapy (GDMT)*
2. Subject with LVEF less than or equal to 35%, sinus rhythm, LBBB with a QRS duration 120 to 149 ms, and NYHA class II, III, or ambulatory IV symptoms on GDMT*
3. Subject with LVEF less than or equal to 35%, sinus rhythm, a non-LBBB pattern with a QRS duration greater than or equal to 150 ms, and NYHA class III/ ambulatory class IV symptoms on GDMT*
4. Subject with atrial fibrillation and LVEF less than or equal to 35% on GDMT* if a) the subject requires ventricular pacing or otherwise meets CRT criteria [listed here] and b) AV nodal ablation or pharmacologic rate control will allow near 100% ventricular pacing with CRT
5. Subject on GDMT* who have LVEF less than or equal to 35% and are undergoing new device placement with anticipated requirement for significant (>40%) ventricular pacing *GDMT = Guideline-directed medical therapy (formerly known as optimal pharmaceutical therapy (OPT)), represents optimal medical therapy as defined by ACCF/ AHA guideline-recommended therapies (primarily Class I)

   * Subject is intended to receive the ACUITY X4 LV lead and RELIANCE 4-FRONT RV lead (optional in Study Phase 1) and BSC CRT-D with quadripolar header as their initial (de novo) cardiac implants
   * Subject is willing and capable of providing informed consent (which can include the use of a legally authorized representative [LAR] for documentation of informed consent) and participating in all testing associated with this investigation at an approved center and at the intervals defined by this protocol
   * Subject is age 18 or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

Subjects who meet any one of the following criteria will be excluded from this clinical study.

* Subject has a known or suspected sensitivity to dexamethasone acetate (DXA)
* Subject has a mechanical tricuspid heart valve
* Subject is enrolled in any other concurrent study, with the exception of local mandatory governmental registries and observational studies/registries* that are not in conflict and do not affect the following:
* Schedule of procedures for the Study (i.e. should not cause additional or missed visits);
* Study outcome (i.e. involve medications that could affect the heart rate of the subject);
* Conduct of the Study per good clinical practice (GCP) / International Organization for Standardization (ISO) 14155:2011/ 21 Code of Federal Regulations (CFR) 812, local regulations
* Subject is currently on the active heart transplant list
* Subject has a documented life expectancy of less than twelve months
* Women of childbearing potential who are or might be pregnant at the time of study enrollment or CRT-D System implant (method of assessment upon physician's discretion)
* Subjects currently requiring chronic dialysis *Sponsors of such studies/registries should be informed and Boston Scientific must be informed by the investigator about the parallel conduct of these projects in the subject and of the project's basic nature. The decision if a desired mandatory governmental registry or observational study/ registry is in conflict with this exclusion criterion is up to the enrolling investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2244 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2020-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suneet Mittal, MD, Principal Investigator — The Valley Hospital; Martin Burke, DO, Principal Investigator — University of Chicago
Locations (96):
- United States (96):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Huntsville Hospital, Huntsville, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Baywood Heart Hospital, Mesa, Arizona
  - Scottsdale Healthcare - Osborn, Scottsdale, Arizona
  - Cardiology Associates of Northeast Arkansas, P.A., Jonesboro, Arkansas
  - Kaiser Permanente, Los Angeles, California
  - USC Medical Center, Los Angeles, California
  - Alta Bates Medical Center, Oakland, California
  - Mercy General Hospital, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Delray Medical Center, Fort Lauderdale, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - West Florida Cardiology Network, LLC, Largo, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Gwinnett Hospital System Inc., Lawrenceville, Georgia
  - University of Chicago, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Porter Memorial Hospital, Dyer, Indiana
  - Lutheran Medical Group, Fort Wayne, Indiana
  - St. Vincent's Hospital, Indianapolis, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Eastern Maine Medical Center, Bangor, Maine
  - Union Memorial Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - St. Joseph Mercy Hospital, Ypsilanti, Michigan
  - St. Mary's Duluth Clinic Regional Heart Center, Duluth, Minnesota
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - Boone Hospital Center, Columbia, Missouri
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Cox Health, Springfield, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Cooper Hospital - University Medical Center, Haddon Heights, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Buffalo General Hospital, Williamsville, New York
  - Mercy Hospital of Buffalo, Catholic Health System, Williamsville, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - OhioHealth Research and Innovation Institute - Riverside Methodist Hospital, Columbus, Ohio
  - Wheeling Hospital Inc., Steubenville, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - PeeDee Cardiology Associates PA, Florence, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Heart Hospital of South Dakota, Sioux Falls, South Dakota
  - Stern Cardiovascular Foundation, Inc., Germantown, Tennessee
  - St. Thomas Research Institute, LLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - Heart Hospital of Austin, Austin, Texas
  - SouthEast Texas Clinical Research Center, Beaumont, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Walnut Hill Medical Center, Dallas, Texas
  - Plaza Medical Center of Fort Worth, Fort Worth, Texas
  - University of Texas Houston Health Science Center, The Woodlands, Texas
  - Trinity Mother Frances Health System, Tyler, Texas
  - Intermountain Medical Center, Murray, Utah
  - Bon Secours Heart & Vascular Institute, Mechanicsville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Cardiovascular Specialist, Richmond, Virginia
  - PeaceHealth St. Joseph Medical Center, Bellingham, Washington
  - Providence Regional Medical Center Everett, Everett, Washington
  - Kootenai Heart Clinics, Spokane, Washington
  - Providence Health & Services - Washington, Spokane, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - Monongalia General Hospital, Morgantown, West Virginia

REFERENCES:
- [Derived] Mittal S, Nair D, Padanilam BJ, Ciuffo A, Gupta N, Gallagher P, Goldner B, Hammill EF, Wold N, Stein K, Burke M. Performance of Anatomically Designed Quadripolar Left Ventricular Leads: Results from the NAVIGATE X4 Clinical Trial. J Cardiovasc Electrophysiol. 2016 Oct;27(10):1199-1205. doi: 10.1111/jce.13044. Epub 2016 Aug 19. PMID 27434039

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were not randomized to received a specific lead.
Groups:
- NAVIGATE X4 Study Participants: All subjects that signed the informed consent were included.
  Subjects consent to undergo an implant procedure to receive at least one study device: ACUITY X4 LV lead, RELIANCE 4-FRONT RV lead. Each subject was allowed to be implanted with both leads.
  ACUITY X4 quadripolar coronary venous lead: The ACUITY X4 leads are intended for chronic left ventricular pacing and sensing. The leads have 3 tip configuration designs (straight tip, short tip spiral, and long tip spiral), which is intended to provide choices for patients with different anatomies.
  RELIANCE 4-FRONT defibrillation lead: The RELIANCE 4-FRONT leads are designed for right-side heart applications within the ventricle, atrium, and superior vena cava. It is intended for permanent sensing, pacing, and defibrillation when used with a compatible ICD or CRT-D.
Period: Overall Study
Arm/Group | NAVIGATE X4 Study Participants
Started | 2244
Implanted/Attempted With a Study Device (2045 with ACUITY X4 and RELIANCE 4-FRONT, 110 with ACUITY X4 only, 45 with RELIANCE 4-FRONT only) | 2200
RELIANCE 4-FRONT Endpoint Population (The first 1544 subjects implanted/attempted with 4-FRONT lead eligible for 4-FRONT endpoints) | 1544 (1507 with active fixation 4-FRONT lead, 37 with passive fixation 4-FRONT lead)
ACUITY X4 Endpoint Population (The first 764 subjects implanted/attempted with ACUITY X4 lead eligible for ACUITY X4 endpoints) | 764 (536 with ACUITY X4 Spiral lead, 228 with ACUITY X4 Straight lead)
Completed | 409 (Follow-up is ongoing. Data as of 5-Feb-2020.)
Not Completed | 1835

BASELINE CHARACTERISTICS:
Groups:
- NAVIGATE X4 Study Participants: All subjects that signed the informed consent were included.
  Subjects consent to undergo an implant procedure to receive an ACUITY X4 LV lead and/or a RELIANCE 4-FRONT RV lead.
  ACUITY X4 quadripolar coronary venous lead: The ACUITY X4 leads are intended for chronic left ventricular pacing and sensing. The leads have 3 tip configuration designs (straight tip, short tip spiral, and long tip spiral), which is intended to provide choices for patients with different anatomies.
  RELIANCE 4-FRONT defibrillation lead: The RELIANCE 4-FRONT leads are designed for right-side heart applications within the ventricle, atrium, and superior vena cava. It is intended for permanent sensing, pacing, and defibrillation when used with a compatible ICD or CRT-D.
Arm/Group | NAVIGATE X4 Study Participants
Number analyzed (Participants) | 2244
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 777
  Male | 1467
Race (NIH/OMB) [Count of Participants; unit: Participants] — Racial and Ethnic Categories and Definitions consistent with those used for National Institutes of Health (NIH) Diversity Programs/Other Reporting Purposes and with the Standards for the Classification of Federal Data on Race and Ethnicity issued by the Office of Management and Budget (OMB).
  Participants
    American Indian or Alaska Native | 0
    Asian | 22
    Native Hawaiian or Other Pacific Islander | 2
    Black or African American | 292
    White | 1791
    More than one race | 8
    Unknown or Not Reported | 129
Region of Enrollment [Number; unit: participants]
  United States | 2244
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: %] | 25.2 (6.5)
QRS duration [Mean (Standard Deviation); unit: milliseconds] — The QRS duration represents the time for ventricular depolarization (activation), starting at the Q wave and ending at the S wave, as measured from an electrocardiogram (ECG). Q waves are inscribed when the initial QRS vector is directed away from the positive electrode. The R wave is the first positive deflection of the QRS complex. The negative deflection after the R wave is the S wave. Population: Measurement not available on 3 subjects
  milliseconds
    number analyzed (Participants) | 2241
    (all) | 153 (22)
New York Heart Association (NYHA) Classification [Count of Participants; unit: Participants] — NYHA Classification of severity of heart failure places subjects in 1 of 4 categories based on how much they are limited during physical activity, based on physician assessment.
  Class I = normal function status, Class II = Slight limitation of functional status, Class III = Marked limitation of functional status, Class IV = Severe limitation of functional status.
  Participants
    Class I | 5
    Class II | 667
    Class III | 1485
    Class IV | 54
    Non-Heart Failure Subject | 6
    Not available | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of ACUITY X4 Spiral Leads Free From Complication Through 6 Months
Description: Lead-related complication-free rate of ACUITY X4 Spiral Leads from implant through 6 months post implant.
Time Frame: Implant through 6 months
Population: This endpoint was limited to the first 536 subjects implanted/attempted with ACUITY X4 Spiral leads
Measure: Number (97.5% Confidence Interval); unit: % of leads free from complication
Groups:
- NAVIGATE X4 Study Participants: Subjects enrolled in the NAVIGATE X4 Study
Arm/Group | NAVIGATE X4 Study Participants
Number analyzed (Participants) | 536
% of leads free from complication | 98.5 [97.0 to NA] — One-sided test was performed with 2.5% alpha. Lower one-sided 97.5% confidence limit was compared to performance goal of 87%. It was pre-specified to only calculate the lower confidence interval.
Statistical Analysis 1: Comparison: NAVIGATE X4 Study Participants; Ho: The Implant through 6-month lead-related complication-free rate ≤ 87%, Ha: The Implant through 6-month lead-related complication-free rate > 87%; Test type: Superiority — Single group test comparison to a performance goal of 87%. Lower one-sided 97.5% confidence limit was compared to the performance goal. If lower confidence limit exceeded performance goal, null hypothesis was rejected; Percent = 98.5, 97.5% CI 1-sided [lower limit 97.0]

2. Primary Outcome: Percentage of ACUITY X4 Straight Leads Free From Complication Through 6 Months
Description: Lead-related complication-free rate of ACUITY X4 Straight Leads from implant through 6 months post implant.
Time Frame: Implant through 6 months
Population: This endpoint was limited to the first 228 subjects implanted/attempted with ACUITY X4 Straight leads
Measure: Number (95% Confidence Interval); unit: % of leads free from complication
Arm/Group | NAVIGATE X4 Study Participants
Number analyzed (Participants) | 228
% of leads free from complication | 96.5 [93.8 to NA] — One-sided test was performed with 5% alpha. Lower one-sided 95% confidence limit was compared to performance goal of 85%. It was pre-specified to only calculate the lower confidence interval.
Statistical Analysis 1: Comparison: NAVIGATE X4 Study Participants; Ho: The Implant through 6-month lead-related complication-free rate ≤ 85%, Ha: The Implant through 6-month lead-related complication-free rate > 85%; Test type: Superiority — Single group test comparison to a performance goal of 85%. Lower one-sided 95% confidence limit was compared to the performance goal. If lower confidence limit exceeded performance goal, null hypothesis was rejected; Percent = 96.5, 95% CI 1-sided [lower limit 93.8]

3. Primary Outcome: Percentage of ACUITY X4 Leads With Acceptable Pacing Capture Thresholds (PCT)
Description: PCT measurements in the programmed configuration were collected at 3 months post-implant. Programmed configuration refers to the pacing configuration that was selected by the physician to provide LV pacing therapy. The percentage of measurements with PCT ≤ 2.5 V were calculated.
Time Frame: Implant through 3 months
Population: Subjects eligible for endpoint analysis included the first 764 subjects implanted/attempted with ACUITY X4 lead. 685 of these 764 had PCT measurements at 3 months and were included in the evaluation.
Measure: Number (97.5% Confidence Interval); unit: % of leads with acceptable threshold
Arm/Group | NAVIGATE X4 Study Participants
Number analyzed (Participants) | 685
% of leads with acceptable threshold | 94.0 [92.0 to NA] — One-sided test was performed with 2.5% alpha. Lower one-sided 97.5% confidence limit was compared to performance goal of 75%. It was pre-specified to only calculate the lower confidence interval.
Statistical Analysis 1: Comparison: NAVIGATE X4 Study Participants; Ho: Percentage of PCT less than or equal to 2.5V ≤ 75%, Ha: Percentage of PCT less than or equal to 2.5V > 75%; Test type: Superiority — Single group test comparison to a performance goal of 75%. Lower one-sided 97.5% confidence limit was compared to the performance goal. If lower confidence limit exceeded performance goal, null hypothesis was rejected; Percent = 94.0, 97.5% CI 1-sided [lower limit 92.0]

4. Primary Outcome: Percentage of ACUITY X4 Spiral Leads With Acceptable Pacing Capture Thresholds (PCT) Using the Best Proximal Electrode
Description: PCT measurements in the in the proximal zone (electrodes 2, 3, 4) were collected at 3 months post-implant. Physician investigators were instructed to use the best proximal electrode (E2, E3 or E4) as the cathode and the RV lead coil or pulse generator as the anode; best was defined as the electrode with the lowest PCT without phrenic nerve stimulation. The percentage of measurements with PCT ≤ 2.5 V were calculated.
Time Frame: 3 months
Population: Subjects eligible for endpoint analysis included the first 536 subjects implanted/attempted with ACUITY X4 Spiral lead. 484 of these 536 had PCT measurements at 3 months and were included in the evaluation.
Measure: Number (97.5% Confidence Interval); unit: % of leads with acceptable threshold
Arm/Group | NAVIGATE X4 Study Participants
Number analyzed (Participants) | 484
% of leads with acceptable threshold | 91.1 [88.2 to NA] — One-sided test was performed with 2.5% alpha. Lower one-sided 97.5% confidence limit was compared to performance goal of 75%.It was pre-specified to only calculate the lower confidence interval.
Statistical Analysis 1: Comparison: NAVIGATE X4 Study Participants; Ho: Percentage of PCT less than or equal to 2.5V ≤ 75%, Ha: Percentage of PCT less than or equal to 2.5V > 75%; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Percent = 91.1, 97.5% CI 1-sided [lower limit 88.2]

5. Primary Outcome: Percentage of RELIANCE 4-FRONT Leads Free From Complication Through 3 Months
Description: Lead-related complication-free rate of RELIANCE 4-FRONT Leads from implant through 3 months post implant.
Time Frame: Implant through 3 months
Population: This endpoint was limited to the first 1544 subjects implanted/attempted with RELIANCE 4-FRONT leads. Data from participants were pooled with data from 334 subjects from 2 other studies for official endpoint analysis. Only data from NAVIGATE X4 are presented here.
Measure: Number (95% Confidence Interval); unit: % of leads free from complication
Arm/Group | NAVIGATE X4 Study Participants
Number analyzed (Participants) | 1544
% of leads free from complication | 98.2 [97.5 to NA] — One-sided test was performed with 5% alpha. Lower one-sided 95% confidence limit was compared to performance goal of 93%. It was pre-specified to only calculate the lower confidence interval.
Statistical Analysis 1: Comparison: NAVIGATE X4 Study Participants; Ho: The Implant through 3-month lead-related complication-free rate ≤ 93%, Ha: The Implant through 3-month lead-related complication-free rate > 93%; Test type: Superiority — Single group test comparison to a performance goal of 93%. Lower one-sided 95% confidence limit was compared to the performance goal. If lower confidence limit exceeded performance goal, null hypothesis was rejected; Percent = 98.2, 95% CI 1-sided [lower limit 97.5]

6. Primary Outcome: Percentage of RELIANCE 4-FRONT Leads Free From Complication From 3 Through 24 Months
Description: Lead-related complication-free rate of RELIANCE 4-FRONT Leads from 3 through 24 months post implant.
Time Frame: 3 months through 24 months
Population: The first 1544 subjects implanted/attempted with RELIANCE 4-FRONT leads were eligible for endpoint analysis. Of these 1544, leads still in service at 3 months were evaluated (n = 1486). Data from participants were pooled with data from subjects from 2 other studies for official endpoint analysis. Only data from NAVIGATE X4 are presented here.
Measure: Number (95% Confidence Interval); unit: % of leads free from complication
Arm/Group | NAVIGATE X4 Study Participants
Number analyzed (Participants) | 1486
% of leads free from complication | 99.3 [98.8 to NA] — One-sided test was performed with 5% alpha. Lower one-sided 95% confidence limit was compared to performance goal of 94%. It was pre-specified to only calculate the lower confidence interval.
Statistical Analysis 1: Comparison: NAVIGATE X4 Study Participants; Ho: The 3- through 24-month lead-related complication-free rate ≤ 94%, Ha: The 3- through 24-month lead-related complication-free rate > 94%; Test type: Superiority — Single group test comparison to a performance goal of 94%. Lower one-sided 95% confidence limit was compared to the performance goal. If lower confidence limit exceeded performance goal, null hypothesis was rejected; Percent = 99.3, 95% CI 1-sided [lower limit 98.8]

7. Primary Outcome: Mean Pacing Capture Threshold (PCT) of RELIANCE 4-FRONT Leads at 3 Months
Description: PCT measurements from RELIANCE 4-FRONT leads were collected at 3 months post-implant. Measurements were performed using 0.5 millisecond pulse width.
Time Frame: Implant through 3 months
Population: Subjects eligible for endpoint analysis included the first 1544 subjects implanted/attempted with RELIANCE 4-FRONT lead. 1432 of these 1544 had PCT measurements at 3 months and were included in the evaluation. Data were pooled with data from subjects from 2 other studies for official endpoint analysis. Only data from NAVIGATE X4 are presented here.
Measure: Mean (95% Confidence Interval); unit: Volts (V)
Arm/Group | NAVIGATE X4 Study Participants
Number analyzed (Participants) | 1432
Volts (V) | 0.56 [NA to 0.58] — One-sided test was performed with 5% alpha. Upper one-sided 95% confidence limit was compared to performance goal of 1.5 Volts. It was pre-specified to only calculate the upper confidence interval.
Statistical Analysis 1: Comparison: NAVIGATE X4 Study Participants; Ho: The 3-month mean PCT ≥ 1.5 Volts, Ha: The 3-month mean PCT < 1.5 Volts; Test type: Superiority — Single group test comparison to a performance goal of 1.5 Volts. Upper one-sided 95% confidence limit was compared to the performance goal. If upper confidence limit was lower than the performance goal, null hypothesis was rejected; Mean = 0.56, 95% CI 1-sided [upper limit 0.58]

8. Secondary Outcome: Mean Sensed Amplitude of ACUITY X4 Spiral Leads at 3 Months
Description: Sensed amplitude measurements from ACUITY X4 Spiral leads were collected at 3 months post-implant.
Time Frame: 3 months
Population: Subjects eligible for endpoint analysis included the first 536 subjects implanted/attempted with ACUITY X4 Spiral lead. 457 of these 536 had sensed amplitude measurements at 3 months and were included in the evaluation.
Measure: Mean (97.5% Confidence Interval); unit: millivolts (mV)
Arm/Group | NAVIGATE X4 Study Participants
Number analyzed (Participants) | 457
millivolts (mV) | 17.4 [16.7 to NA] — One-sided test was performed with 2.5% alpha. Lower one-sided 97.5% confidence limit was compared to performance goal of 3 mV. It was pre-specified to only calculate the lower confidence interval.
Statistical Analysis 1: Comparison: NAVIGATE X4 Study Participants; Ho: The 3-month mean sensed amplitude ≤ 3 mV, Ha: The 3-month mean sensed amplitude > 3 mV; Test type: Superiority — Single group test comparison to a performance goal of 3 mV. Lower one-sided 95% confidence limit was compared to the performance goal. If lower confidence limit was greater than the performance goal, null hypothesis was rejected; Mean = 17.4, 95% CI 1-sided [lower limit 16.7]

9. Secondary Outcome: Mean Sensed Amplitude of ACUITY X4 Straight Leads at 3 Months
Description: Sensed amplitude measurements from ACUITY X4 Straight leads were collected at 3 months post-implant.
Time Frame: 3 months
Population: Subjects eligible for endpoint analysis included the first 228 subjects implanted/attempted with ACUITY X4 Straight lead. 189 of these 228 had sensed amplitude measurements at 3 months and were included in the evaluation.
Measure: Mean (97.5% Confidence Interval); unit: millivolts (mV)
Arm/Group | NAVIGATE X4 Study Participants
Number analyzed (Participants) | 189
millivolts (mV) | 16.1 [15.1 to NA] — One-sided test was performed with 2.5% alpha. Lower one-sided 97.5% confidence limit was compared to performance goal of 85%. It was pre-specified to only calculate the lower confidence interval.
Statistical Analysis 1: Comparison: NAVIGATE X4 Study Participants; Ho: The 3-month mean sensed amplitude ≤ 3 mV, Ha: The 3-month mean sensed amplitude > 3 mV; Test type: Superiority — [test comment as in outcome 8, analysis 1]; Mean = 16.1, 97.5% CI 1-sided [lower limit 15.1]

10. Secondary Outcome: Mean Pacing Impedance of ACUITY X4 Spiral Leads at 3 Months
Description: Pacing impedance measurements from ACUITY X4 Spiral leads were collected at 3 months post-implant.
Time Frame: 3 months
Population: Subjects eligible for endpoint analysis included the first 536 subjects implanted/attempted with ACUITY X4 Spiral lead. 482 of these 536 had pacing impedance measurements at 3 months and were included in the evaluation.
Measure: Mean (97.5% Confidence Interval); unit: ohms
Arm/Group | NAVIGATE X4 Study Participants
Number analyzed (Participants) | 482
ohms | 776 [753 to NA] — One-sided test was performed with 2.5% alpha. Lower one-sided 97.5% confidence limit was compared to performance goal of 300 ohms. It was pre-specified to only calculate the lower confidence interval.
Statistical Analysis 1: Comparison: NAVIGATE X4 Study Participants; Ho: The 3-month mean pacing impedance ≤ 300 ohms, Ha: The 3-month mean pacing impedance > 300 ohms; Test type: Superiority — Single group test comparison to a performance goal of 300 ohms. Lower one-sided 95% confidence limit was compared to the performance goal. If lower confidence limit was greater than the performance goal, null hypothesis was rejected; Mean = 776, 97.5% CI 1-sided [lower limit 753]

11. Secondary Outcome: Mean Pacing Impedance ACUITY X4 Straight Leads at 3 Months
Description: Pacing impedance measurements from ACUITY X4 Straight leads were collected at 3 months post-implant.
Time Frame: 3 months
Population: Subjects eligible for endpoint analysis included the first 228 subjects implanted/attempted with ACUITY X4 Straight lead. 202 of these 228 had pacing impedance measurements at 3 months and were included in the evaluation.
Measure: Mean (97.5% Confidence Interval); unit: ohms
Arm/Group | NAVIGATE X4 Study Participants
Number analyzed (Participants) | 202
ohms | 805 [763 to NA] — One-sided test was performed with 2.5% alpha. Lower one-sided 97.5% confidence limit was compared to performance goal of 300 ohms. It was pre-specified to only calculate the lower confidence interval.
Statistical Analysis 1: Comparison: NAVIGATE X4 Study Participants; Ho: The 3-month mean pacing impedance ≤ 300 ohms, Ha: The 3-month mean pacing impedance > 300 ohms; Test type: Superiority — [test comment as in outcome 10, analysis 1]; Mean = 805, 97.5% CI 1-sided [lower limit 763]

12. Secondary Outcome: Mean Detection Time of Induced Ventricular Tachycardia / Ventricular Fibrillation (VT/VF) Episodes Using RELIANCE 4-FRONT Leads
Description: The mean detection time, in seconds, of induced VT/VF episodes occurring within 30 days of implant were evaluated. Subjects were required to implanted with RELIANCE 4-FRONT leads to be evaluated.
Time Frame: Within 30 days of implant
Population: Subjects eligible for endpoint analysis included the first 1544 subjects implanted/attempted with RELIANCE 4-FRONT lead. 557 of these 1544 had induced VT/VF episodes within 30 days of implant with detection time data and were included in the evaluation.
Measure: Number (95% Confidence Interval); unit: seconds
Arm/Group | NAVIGATE X4 Study Participants
Number analyzed (Participants) | 557
seconds | 3.14 [NA to 3.2] — One-sided test was performed with 5% alpha. Upper one-sided 95% confidence limit was compared to performance goal of 4.5 seconds. It was pre-specified to only calculate the upper confidence interval.
Statistical Analysis 1: Comparison: NAVIGATE X4 Study Participants; Ho: The mean detection time ≥ 4.5 seconds, Ha: The mean detection time < 4.5 seconds; Test type: Superiority — Single group test comparison to a performance goal of 4.5 seconds. Upper one-sided 95% confidence limit was compared to the performance goal. If upper confidence limit was lower than the performance goal, null hypothesis was rejected; Mean = 3.14, 95% CI 1-sided [upper limit 3.20]

13. Secondary Outcome: Mean Sensed Amplitude of RELIANCE 4-FRONT Leads at 3 Months
Description: Sensed amplitude measurements from RELIANCE 4-FRONT leads were collected at 3 months post-implant.
Time Frame: 3 months
Population: Subjects eligible for endpoint analysis included the first 1544 subjects implanted/attempted with RELIANCE 4-FRONT lead. 1374 of these 1544 had sensed amplitude at 3 months and were included in the evaluation. Data were pooled with data from subjects from 2 other studies for official endpoint analysis. Only data from NAVIGATE X4 are presented here.
Measure: Mean (95% Confidence Interval); unit: millivolts (mV)
Arm/Group | NAVIGATE X4 Study Participants
Number analyzed (Participants) | 1374
millivolts (mV) | 18.3 [17.9 to NA] — One-sided test was performed with 5% alpha. Lower one-sided 95% confidence limit was compared to performance goal of 5 mV seconds. It was pre-specified to only calculate the lower confidence interval.
Statistical Analysis 1: Comparison: NAVIGATE X4 Study Participants; Ho: The 3-month mean sensed amplitude ≤ 5 mV, Ha: The 3-month mean sensed amplitude > 5 mV; Test type: Superiority — Single group test comparison to a performance goal of 5 mV. Lower one-sided 95% confidence limit was compared to the performance goal. If lower confidence limit was greater than the performance goal, null hypothesis was rejected; Mean = 18.3, 95% CI 1-sided [lower limit 6.2]

14. Secondary Outcome: Mean Pacing Impedance of RELIANCE 4-FRONT Active Fixation Leads at 3 Months
Description: Pacing impedance measurements from RELIANCE 4-FRONT Active Fixation leads were collected at 3 months post-implant.
Time Frame: 3 months
Population: Subjects eligible for analysis included the first 1507 subjects implanted/attempted with RELIANCE 4-FRONT active fixation lead. 1402 of these 1544 had pacing impedance measurements at 3 months and were included in the evaluation. Data were pooled with 2 other studies for official endpoint analysis. Only data from NAVIGATE X4 are presented here.
Measure: Mean (90% Confidence Interval); unit: ohms
Arm/Group | NAVIGATE X4 Study Participants
Number analyzed (Participants) | 1402
ohms | 468 [463 to 472]
Statistical Analysis 1: Comparison: NAVIGATE X4 Study Participants; Ho: Pacing impedance ≤ 300 Ω or pacing impedance ≥ 1200 Ω, Ha: 300 Ω < Pacing impedance < 1200 Ω; Test type: Other — Two one-sided tests (TOST) were performed; Mean = 468, 90% CI 2-sided [463 to 472]

15. Secondary Outcome: Mean Pacing Impedance of RELIANCE 4-FRONT Passive Fixation Leads at 3 Months
Description: Pacing impedance measurements from RELIANCE 4-FRONT Passive Fixation leads were collected at 3 months post-implant.
Time Frame: 3 months
Population: Subjects eligible for analysis included the first 37 subjects implanted/attempted with RELIANCE 4-FRONT passive fixation lead. 36 of these 37 had pacing impedance measurements at 3 months and were included in the evaluation. Data were pooled with 2 other studies for official endpoint analysis. Only data from NAVIGATE X4 are presented here.
Measure: Mean (90% Confidence Interval); unit: ohms
Groups:
- RELIANCE 4-FRONT LEAD: RELIANCE 4-FRONT Endpoint Population
Arm/Group | RELIANCE 4-FRONT LEAD
Number analyzed (Participants) | 36
ohms | 702 [659 to 744]
Statistical Analysis 1: Comparison: RELIANCE 4-FRONT LEAD; Ho: Pacing impedance ≤ 300 Ω or pacing impedance ≥ 1200 Ω, Ha: 300 Ω < Pacing impedance < 1200 Ω; Test type: Other — Two one-sided tests (TOST) were performed; Mean = 702, 90% CI 2-sided [659 to 744]

16. Secondary Outcome: Percentage of Successfully Converted Induced Ventricular Tachycardia / Ventricular Fibrillation (VT/VF) Episodes Using RELIANCE 4-FRONT Leads
Description: Ventricular Tachyarrhythmia (VT/VF) Shock Conversion Efficacy, analyzed within 30 days of implant
Time Frame: Within 30 days of implant
Population: Subjects eligible for endpoint analysis included the first 1544 subjects implanted/attempted with RELIANCE 4-FRONT lead. 560 of these 1544 had induced VT/VF episodes within 30 days of implant that were included in the evaluation.
Measure: Number (95% Confidence Interval); unit: % of induced episodes
Arm/Group | NAVIGATE X4 Study Participants
Number analyzed (Participants) | 560
% of induced episodes | 99.5 [98.4 to NA] — One-sided test was performed with 5% alpha. Lower one-sided 95% confidence limit was compared to performance goal of 93%. It was pre-specified to only calculate the lower confidence interval.
Statistical Analysis 1: Comparison: NAVIGATE X4 Study Participants; Ho: Percent of successful conversion ≤ 93%, Ha: Percent of successful conversion > 93%; Test type: Superiority — Single group test comparison to a performance goal of 93%. Lower one-sided 95% confidence limit was compared to the performance goal. If lower confidence limit was greater than the performance goal, null hypothesis was rejected; Percent = 99.5, 95% CI 1-sided [lower limit 98.4]

ADVERSE EVENTS:
Time Frame: Entire follow-up: implant through 5 years post-implant (median participant follow-up = 4.3 years).
Description: All adverse events (serious/non-serious, related/unrelated to device) were to be reported to Boston Scientific by the investigational sites. All-cause mortality evaluated in all enrolled participants (N = 2244). Adverse events evaluated in participants implanted or attempted with ACUITY X4 and/or RELIANCE 4-FRONT (N = 2200).
Groups:
- NAVIGATE X4 Study Participants: All-cause mortality evaluated in all enrolled participants (N = 2244). Adverse events evaluated in participants implanted or attempted with ACUITY X4 and/or RELIANCE 4-FRONT (N = 2200). Adverse events were not collected based on the lead implanted in the subject. All subjects were implanted or attempted with a CRT-D, Individual adverse event categories evaluated in participants at risk for that event category (2007 implanted/attempted with RA lead, 2090 with 4-FRONT, 2199 with any RV lead, 2162 with ACUITY X4, 2182 with any LV lead, 2019 with ACUITY X4 and/or 4-FRONT, 2019 with any lead).
Arm/Group | NAVIGATE X4 Study Participants
All-Cause Mortality (participants affected / at risk) | 491/2244
Serious Adverse Events (participants affected / at risk) | 1539/2200
Other Adverse Events (participants affected / at risk) | 1768/2200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | NAVIGATE X4 Study Participants (N=2200)
Cardiovascular - Heart Failure (Cardiac disorders) | 620 (1256)
Cardiovascular - Non-Heart Failure (Cardiac disorders) | 829 (1431)
Non-Cardiovascular (General disorders) | 1043 (2581)
Pulse Generator (Product Issues) | 74 (80)
RA Lead (Product Issues) | 28/2007 (29)
RV Lead - Related to RELIANCE 4-FRONT (Product Issues) | 45/2090 (46)
RV Lead - Unrelated to / Not caused by RELIANCE 4-FRONT (Product Issues) | 6/2199 (6)
LV Lead - Related to ACUITY X4 (Product Issues) | 24/2162 (24)
LV Lead - Unrelated to / Not caused by ACUITY X4 (Product Issues) | 9/2182 (9)
RV & LV Lead - Related to both RELIANCE 4-FRONT and ACUITY X4 (Product Issues) | 3/2109 (3)
Lead - Other (Product Issues) | 16/2019 (17)
Procedure-related (Surgical and medical procedures) | 107 (117)
Unclassified (Investigations) | 5 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | NAVIGATE X4 Study Participants (N=2200)
Cardiovascular - Heart Failure (Cardiac disorders) | 543 (838)
Cardiovascular - Non-Heart Failure (Cardiac disorders) | 1105 (2358)
Non-Cardiovascular (General disorders) | 1341 (5430)
Pulse Generator (Product Issues) | 262 (328)
RA Lead (Product Issues) | 43/2007 (47)
RV Lead - Related to RELIANCE 4-FRONT (Product Issues) | 41/2090 (46)
RV Lead - Unrelated to / Not caused by RELIANCE 4-FRONT (Product Issues) | 4/2199 (4)
LV Lead - Related to ACUITY X4 (Product Issues) | 271/2162 (322)
LV Lead - Unrelated to / Not caused by ACUITY X4 (Product Issues) | 9/2182 (9)
RV & LV Lead - Related to both RELIANCE 4-FRONT and ACUITY X4 (Product Issues) | 8/2109 (8)
Lead - Other (Product Issues) | 6/2109 (6)
Procedure-related (Surgical and medical procedures) | 297 (350)
Unclassified (Investigations) | 8 (9)

LIMITATIONS AND CAVEATS:
Data as of 5-Feb-2020. Follow-up is ongoing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-02-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT02071173/SAP_000.pdf
  • Study Protocol (2013-12-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT02071173/Prot_001.pdf